CLINICAL TRIAL: NCT02466880
Title: Intervention for Diabetes With Education, Advancement and Support (IDEAS) Study
Brief Title: Intervention for Diabetes With Education, Advancement and Support
Acronym: IDEAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: MOSTI Malaysia (Unknown)
Responsible Party: Principal Investigator, Shaun Lee Wen Huey, Senior Lecturer, Monash University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IDEAS001
Record Dates: First submitted 2015-06-02; First posted 2015-06-09 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus
Keywords: Type 2; NIDDM
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine (Experimental): Diabetes education and support via telemedicine
  Interventions: Device: Telemedicine
- Usual care (Active Comparator): Diabetes education and support in person
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Telemedicine — A diabetes self-management and education program delivered via telemedicine
  Arms: Telemedicine
Other: Usual care — A 15-30 minute diabetes self-management session. Continued care, as usual, from their primary care provider throughout duration of active 12 month intervention period.
  Arms: Usual care

SUMMARY:
This study aims to evaluate a culturally appropriate, low cost and sustainable management plan for patients with type 2 diabetes mellitus (T2DM). Various randomized controlled trials confirmed that T2DM can be delayed with lifestyle intervention and programmes which promote improvements in diet, increased physical activity and weight loss. Translation of lifestyle intervention to real-life settings however remains a major challenge.

The investigators therefore propose a diabetes management trial for T2DM patients using telemedicine. This project's innovations include the use of information technology to deliver messages to the physicians while similarly involving family members of diabetics to manage the patient's condition collectively. This creates a sense of well-being, empowering the individual as well as the community to be responsible for their own health and well-being

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes diagnosed by a physician at least six months prior to study enrollment
* HbA1c of > 7.5% but less than 11.0% within the most recent 3 months
* Access to internet and an e-mail address , or access to a smartphone with 3G services
* Not pregnant or history of heart diseases, serious illness, cancer diagnosis or any other conditions that can impede participation

Exclusion Criteria:

* Unable or unwilling to give informed consent or communicate with local study staff
* Current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder
* Hospitalization for depression in past six months
* Plans to relocate to an area or travel plans that do not permit full participation in the study
* Lack of support from primary health care provider or family members
* History of bariatric surgery, small bowel resection, or extensive bowel resection
* Currently pregnant or nursing
* Cancer: requiring treatment in the past five years, except for non-melanoma skin cancers or cancers that have clearly been cured or in the opinion of the investigator carry an excellent prognosis (e.g., Stage 1 cervical cancer)
* Cardiovascular disease (heart attack or procedure within the past three months or participation in a cardiac rehabilitation program within last three months, stroke or history/treatment for transient ischemic attacks in the past three months, or documented history of pulmonary embolus in past six months)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-04; Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c | 3 months, 6 months, 12 months

SECONDARY OUTCOMES:
Change in Quality of life - Measured with EQ5D | 3 months, 6 months, 12 months
Change in Blood pressure | 3 months, 6 months, 12 months
Change in Weight | 3 months, 6 months, 12 months
Cost effectiveness and cost utility | 1 year
  The objectives are to compare the results of the study to that of usual care in patients with type 2 diabetes in terms of cost, cost-effectiveness and cost utility of these two strategies.
Change in Cholesterol | 3 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik Kesihatan Pandamaran, Klang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Publication in peer review journal

REFERENCES:
- [Derived] Lee JY, Chan CKY, Chua SS, Paraidathathu T, Lee KK, Tan CSS, Nasir N, Lee SWH. Using telemedicine to support care for people with type 2 diabetes mellitus: a qualitative analysis of patients' perspectives. BMJ Open. 2019 Oct 22;9(10):e026575. doi: 10.1136/bmjopen-2018-026575. PMID 31640990
- [Derived] Lee JY, Chan CKY, Chua SS, Ng CJ, Paraidathathu T, Lee KKC, Lee SWH. Telemonitoring and Team-Based Management of Glycemic Control on People with Type 2 Diabetes: a Cluster-Randomized Controlled Trial. J Gen Intern Med. 2020 Jan;35(1):87-94. doi: 10.1007/s11606-019-05316-9. Epub 2019 Sep 11. PMID 31512187
- [Derived] Lee JY, Chan CK, Chua SS, Ng CJ, Paraidathathu T, Lee KK, Lee SW. Intervention for Diabetes with Education, Advancement and Support (IDEAS) study: protocol for a cluster randomised controlled trial. BMC Health Serv Res. 2016 Sep 29;16(1):524. doi: 10.1186/s12913-016-1782-y. PMID 27683021